CLINICAL TRIAL: NCT00493116
Title: A Multi-Centre, Open Label Study to Investigate the Recovery of IFN-beta Efficacy in Relapsing-Remitting Multiple Sclerosis Patients With Neutralising IFN-beta Antibodies and Reduced Bioavailability
Brief Title: Is IFN-beta Treatment in MS Useful After a Washout Period in Patients With Neutralizing Antibodies to Interferon Beta
Acronym: RENeu
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUS-8001
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2011-07

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: recovery of efficacy; MxA protein; neutralizing antibodies; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1a; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Interferon-beta-1a; Drug: methylprednisolone

INTERVENTIONS:
Drug: Interferon-beta-1a — dosage and frequency as per Biogen Idec protocol
  Other Names: Avonex
Drug: methylprednisolone — dosage and frequency as per Biogen Idec protocol

SUMMARY:
This study is to find out if Interferon-beta (IFN-beta) can recover its effectiveness after a washout period in patients with Multiple Sclerosis who have previously developed neutralizing antibodies to Interferon-Beta

DETAILED DESCRIPTION:
This is an explorative multi-centre, open label, non-comparative trial investigating whether it is possible to recover IFN-beta efficacy in breakthrough relapsing-remitting multiple sclerosis patients with high titres of neutralizing IFN-beta antibodies.

Prior to enrollment, treated MS subjects must have been on interferon-beta-1a or interferon-beta-1b for a minimum of 12 months and have reduced bioavailability as defined by the relative expression of MxA mRNA/GAPDH.

Subjects will complete a washout period with concurrent methylprednisolone 500mg PO daily for 3 days every month until they become Neutralizing Antibody negative. Subjects will then be challenged with AVONEX 30mcg IM weekly. Bioavailability will be measured every three months to determine return of biological activity. Clinical and MRI parameters, safety and tolerability will be compared to baseline to determine efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Must have been receiving interferon-beta-1a or interferon-beta-1b for a minimum of 12 consecutive months prior to enrollment
* Relapsing-Remitting Multiple Sclerosis according to Poser or McDonald criteria
* EDSS score of 6 or less
* NAB titre >or equal to 20 via CPE assay or >or equal to 100 via MxA Protein assay measured at least 24 hours after last interferon-beta injection on two consecutive tests at least 3 months apart
* Reduced bioavailability (relative expression of MxA mRNA/GAPDH

Exclusion Criteria:

* History of severe allergic or anaphylactic reaction to human albumin, to any interferon, Methylprednisolone or to any other component of study drugs
* Clinically significant systemic illness
* History of poorly controlled hypertension, diabetes, or osteoporosis
* History of uncontrolled seizures within 3 months of enrollment
* History of Depression or suicidal ideation within 3 months of enrollment
* Serious local infection (abscess or cellulitis) or systemic infection within 8 weeks of study
* abnormal screening blood tests

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2003-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
return of bioavailability of AVONEX (interferon-beta-1a) as measured by induction of MxA mRNA | screening and every 3 months from month 6 to month 27

SECONDARY OUTCOMES:
Proportion of patients becoming neutralizing antibody negative | screening and every 3 months from month 3 to month 27
proportion of patients becoming neutralizing antibody positive after treatment with AVONEX | at baseline and every three months
proportion of patents relapse free | months 6, 12, 18 and 24
total relapses | 27 months
proportion of patients with an increase in EDSS of 1 point | screening, 3, 9, 15, 21, and 27 months
Brain atrophy and cumulative number of enlarging T2 lesions on MRI | months 0, 12, and 27

CONTACTS AND LOCATIONS:
Locations (2):
- Coordinating Research Site, NSW, Australia
- Research Site, Hamilton, New Zealand